CLINICAL TRIAL: NCT00176124
Title: Leukocyte Depletion of Autologous Whole Blood: Impact on Perioperative Infection Rate and Length of Hospital Stay for Hip Arthroplasty Patients
Brief Title: Leukocyte Depletion of Autologous Whole Blood
Acronym: LDAWB-2001
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: Philipps University Marburg (Other)
Responsible Party: Thomas Frietsch, MD PhD, University of Heidelberg
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UniKlinMa-TF-2001-1; ISRCTN 99578441
Record Dates: First submitted 2005-09-11; First posted 2005-09-15 (Estimated); Last update posted 2008-06-10 (Estimated); Status verified 2008-06

CONDITIONS: Infection; Bacterial Infection; Sepsis
Keywords: leukocyte depletion, autologous transfusion,; infection; bacterial infection; sepsis, antibiotics
MeSH Terms: conditions — Infections; Bacterial Infections; Sepsis | interventions — Leukocyte Reduction Procedures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): storage and transfusion of autologous whole blood without leukocyte depletion : Control group
  Interventions: Procedure: leukocyte depletion of whole blood
- 2 (Experimental): storage and transfusion of leukocyte depleted autologous whole blood : leukocyte depletion group
  Interventions: Procedure: leukocyte depletion of whole blood; Other: Leukocyte filtration/Depletion

INTERVENTIONS:
Procedure: leukocyte depletion of whole blood
Other: Leukocyte filtration/Depletion — leukocyte depletion filters as used routinely: filters (prestorage) inherent to the blood bag sets by gravity force following storage on cold plate for 2 hours
  Other Names: Fresenius leukocyte depletion whole blood filters
  Arms: 2

SUMMARY:
Leukocyte depletion of autologous whole blood prior to storage does not reduce infection rate (wound, urinary tract, other), use of antibiotic treatment and length of hospital stay but may increase retransfusion perioperatively during hip arthroplasty and allogenic transfusion rate

DETAILED DESCRIPTION:
Informed Consent Form:

Prior to the first blood donation, in- and exclusion criteria should be tested. Then the patient is to inform by the investigator about the studies aim and participation conditions such as methods, risks, assurance, data security, etc. The patient and the investigator should sign the informed consent form.

Randomization:

If all inclusion criteria are well given and exclusion criteria are absent, the patient could be enrolled and randomized, prior to the first PAD. Enrollment is parallel in all centers until the final number of 1088 is reached. Breaking the seal of the provided randomization envelope with computerized randomization codes completes randomization. Time and date should be noted.

Blinding:

Randomization is done by the investigator, which should manage the blood donation. The blood bags after inline leukocyte depletion prior to storage do not look different from not depleted bags and are labeled only with the patient's identity and the subjects ID. The allocation to the group is to keep secret from patient, surgeon and anesthesiologist.

Treatment:

A PAD:

Group 1 Preoperative Donation of multiple units ( more than 2) 450 mL autologous whole blood and storage without leukocyte depletion Usual criteria and methods of PAD are used according to regional guidelines of blood donations in the respective center.

Group 2 Preoperative Donation of multiple units (more than 2) 450 mL autologous whole blood and storage following leukocyte depletion 2 to 4 hours after whole blood donations, the whole blood bags should be in-line filtered by the use of leukocyte filtration sets (provided by Pall Medical Company). Storage as in group 1 at 4 degree C in a blood fridge.

A as proposal, the Mannheim concept reveals a 95 percent security in avoidance of allogenic transfusions for a blood loss of 20-25 ml per kg body weight: Intended are 3 donations in weekly intervals. If Hb plasma con-tent decreases below 11 g/dL, the donation will be postponed to the fol-lowing week. Surgery is at the fifth week after the first donation.

B Anesthesia and Surgery:

As usual in the center, and without a difference between the two groups anesthesia and surgery should be performed under following aspects:

* At hospital admission, the actual history should be taken, study measures (Appendix 1) and screening laboratory should be withdrawn prior to anesthesia to compute the infection risk assessment of the respective patient 13.
* Both general and regional (spinal or epidural anesthesia) can be performed
* Normothermia of the patients is essential to the infection rate, hypothermia increases the infection rate by every degree! The intra- and postoperative core temperature range will be requested.
* Circulatory monitoring should be performed according to the centers conventions. Monitoring with a 5 channel ECG is suggested. Normovolemia is essential because hypovolemia is related to increased infection rate by hypoperfusion of the wound14-16. Therefore, a central venous catheter is useful but not obligatory, but urine output is required since it is a more sensitive volume indicator in absence of significant heart and renal failure (and common practice in hip surgery). An arterial line is not obligatory required.
* Bladder catheter (Urine production more than 1ml/kg KG/h)
* Cell Savers and hemodilution (iso- or hypervolemic) are not accepted.
* Blood loss is to calculate carefully by subtracting rinsing from suction volumes and weighing sponges and drapes intraoperatively. Postoperatively the drainage volumes are sufficient if not massive expansion of thighs or hip occurs ( however, this should be noted as AE).
* In the case that allogenic transfusion is required additionally, this should be leukodepleted.
* Intra- und postoperative transfusion trigger are similar for autologous and allogenic transfusion:
* Hb greater than 8,5 plus minus 0,5
* HF over 100 plusminus 10 /min or 35% above base line
* MAP below 60 plusminus 5 mmHg or 35% below base line
* Stenocardia, chest pain
* ST-segment changes greater than 0,2 ms

Further documentation of

* ASA
* sex
* weight
* height
* Anesthesia duration
* OP-duration
* Blood loss(intra- and postoperatively)
* Lowest diastole. RR intraoperatively as well as postoperatively POD 0
* Time of transfusions
* Time of urine catheter withdrawal Infection-Monitoring

Parameter:

• Skin inspection

Criteria of wound infection:

* secretion clear or pus,
* pos. bacterial culture,
* erythema

  * Urine culture if indicated by sediment (at withdrawl of bladder cathe-ter, discolored urine or fever)
  * Blood culture (if fever above 39°C after POD2)
  * Tracheal secretion (if expectoration is prutride or radiological indica-tion of bronchopneumonia)
  * Antibiotic treatment, duration, amounts, multidrug use

Woundhealing and the occurrence of infections were classified with the ASEPSIS score: Of influence is the duration of antibiotic treatment, drainage of pus, wound de-bridements, erythema, involvement of deeper tissue layers, identification of bacteria, LOS above 14 days 17.

Infection Definition

Occurrence of any infection is defined as

* Elevation of patient's temperature/fever above 38°C on POD 3 or later or
* Leukocytosis above the cut off point (generated for every individual subject )or
* BSG / CRP above the cut off point (generated for every individual subject ) or
* Isolation of bacteria from any fluid including pus or
* Abscess (verificated by surgical drainage or ultrasonographically guided aspiration of pus ) or
* Arthritis by local clinical symptoms and surgical drainage

Wound infection is assessed by the ASEPSIS score

Urinary tract infection is defined as

* new isolated occurrence of leukocytosis, and/or nitrite, and/or protein or
* isolation of bacteria more than 10 000/µl (sediment) or
* growth of more than 100 000 colonies of a single organism in the culture

Respiratory airway infection is defined as

* positive x-ray (chest infiltrate) and fever or
* dyspnea or cough or purulent sputum and fever or
* isolation of bacteria in tracheal secretion (only intubated subjects) and fever

Septicemia is defined as

• clinical symptoms and positive blood culture

ELIGIBILITY:
Inclusion Criteria:

* • ASA I-III,

  * Age 18-85 years,
  * Body weight 50-125 kg
  * If female, with either a history of an accepted method of anticonception for at least 3 month prior and 1 month following the termination of the study or climacteric or with a negative betA- HCG-Test in urine or serum.
  * Preoperative blood donation of at least 2 units (450mL whole blood)
  * Preoperative hemoglobin level > 10 mg/dL
  * Able and willing to sign informed consent

Exclusion Criteria:

* Subjects with a contraindication for preoperative blood donation (PAD) (in 12, PP 36-43).

  * systemic infection
  * acute bacterial or viral diseases
  * anemia (Hb > 11g/dL)
  * myocardial infarction within the past 6 month,
  * instable angina pectoris
  * vascular stenosis (i.e. of the coronary or internal carotid arteries)
  * hemodynamic relevant valvular stenosis
  * heart failure > NYHA II
  * history of strokes or TIA
  * steroid therapy,
  * immune deficiency,
  * hematological or endocrinological disease,
  * coagulopathy,
  * history of organ transplantation,
  * simultaneous participation in a second study
  * pregnancy
  * membership at Jehovah's Witnesses
  * intended use of a cell saver

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1089 (Actual)
Dates: Start 2001-04; Primary Completion 2005-04 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Comparison of infection rate (wound, urinary tract, other), use of antibiotic treatment and length of hospital stay | 90 days

SECONDARY OUTCOMES:
Blood loss and transfusion rate | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Frietsch, MD, PhD, Study Chair — Clinic of Anesthesiology and Critical Care Medicine, Faculty of Clinical Medicine Mannheim, University of Heidelberg
Locations (3):
- Germany (3):
  - Clinic of Anesthesiology and Critical Care Medicine, Faculty of Clinical Medicine MAnnheim, University of Heidelberg, Germany, Mannheim, Baden-Wurttemberg
  - Klinikum Garmisch Partenkirchen, Garmisch-Partenkirchen, Bavaria
  - Institute of Transfusion Medicine and Hemostasiology, University of MArburg, Marburg

REFERENCES:
- [Background] Byrne DJ, Malek MM, Davey PG, Cuschieri A. Postoperative wound scoring. Biomed Pharmacother. 1989;43(9):669-73. doi: 10.1016/0753-3322(89)90085-1. PMID 2696565
- [Background] Frietsch T, Fessler H, Kirschfink M, Nebe T, Waschke KF, Lorentz A. Immune response to autologous transfusion in healthy volunteers: WB versus packed RBCs and FFP. Transfusion. 2001 Apr;41(4):470-6. doi: 10.1046/j.1537-2995.2001.41040470.x. PMID 11316896
- [Background] Frietsch T, Krombholz K, Tolksdorf B, Nebe T, Segiet W, Lorentz A. Cellular immune response to autologous blood transfusion in hip arthroplasty: whole blood versus buffy coat-poor packed red cells and fresh-frozen plasma. Vox Sang. 2001 Oct;81(3):187-93. doi: 10.1046/j.1423-0410.2001.00107.x. PMID 11703863
- [Background] Lorentz A, Osswald PM, Schilling M, Jani L. [A comparison of autologous transfusion procedures in hip surgery]. Anaesthesist. 1991 Apr;40(4):205-13. German. PMID 2058822
- [Background] Tolksdorf B, Frietsch T, Quintel M, Kirschfink M, Becker P, Lorentz A. Humoral immune response to autologous blood transfusion in hip surgery: whole blood versus packed red cells and plasma. Vox Sang. 2001 Oct;81(3):180-6. doi: 10.1046/j.1423-0410.2001.00106.x. PMID 11703862
- [Background] Frietsch T, Lorentz A. Predonation of autologous blood is jeopardized by new regulations. Eur J Anaesthesiol. 2001 Oct;18(10):629-31. doi: 10.1046/j.1365-2346.2001.00997.x. No abstract available. PMID 11553239